CLINICAL TRIAL: NCT05790954
Title: The Effect of Pre-Cesarean Section Guided Imagery on Preoperative Anxiety, Fear and Physiological Parameters
Brief Title: The Effect of Pre-Cesarean Section Guided Imagery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menekşe Nazlı AKER (Other)
Responsible Party: Sponsor-Investigator, Menekşe Nazlı AKER, Assist. Prof., Ankara University
Organization: Ankara University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 15149
Record Dates: First submitted 2023-03-17; First posted 2023-03-30 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Cesarean Section
MeSH Terms: interventions — Imagery, Psychotherapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guided imagery Group (Experimental)
  Interventions: Other: Guided imagery
- Control Group (No Intervention)

INTERVENTIONS:
Other: Guided imagery — Three days before the cesarean section, the participants will be given a guided imagery audio recording and will be asked to listen to it before going to bed every evening until the day of the cesarean section. On the morning of the cesarean section, after the patient is prepared, the guided imagery audio recording will be played again.
  Arms: Guided imagery Group

SUMMARY:
The aim of this study is to evaluate the effect of guided imagery applied before cesarean section on preoperative anxiety, fear and physiological parameters.

The study will be carried out in two different groups. The practice will start with meeting the women 3 days before cesarean section. After the women are evaluated in terms of eligibility criteria for the research, the women who are eligible will be informed about the research and written informed consent will be obtained from the women who accept. The random distribution of women to the study groups will be carried out random. The following applications will be made to the groups.

ELIGIBILITY:
Inclusion Criteria:

* planned cesarean section
* Single birth
* giving birth at term
* No hearing problems
* Agreeing to participate in the research and obtaining written permission,

Exclusion Criteria:

* Emergency cesarean section due to a health problem of the mother or baby
* Not completing the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-03-27 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Change in anxiety | Three days before the cesarean section, Fifteen minutes after preparation for cesarean section
  The State-Trait Anxiety Inventory-S consist of 20 items with four points likert scales, each (not at all, somewhat, moderately so, very much so). Scores thus range between 20, indicating a low level of anxiety and 80, indicating a high level.
Change in Surgical Fear | Three days before the cesarean section, Fifteen minutes after preparation for cesarean section
  Surgical Fear Questionnaire has been developed to determine the level of fear of patients who will undergo electrical surgery for the short and long -term results of surgical operation. The scale is a scales of 11 Likertes, which consist of 8 items, scored between 0-10. Each item 0 is scored as "I'm at all scared", 10 "I'm very scared". The total score of the scale is 0-80. The high score states that surgical fear is high.

SECONDARY OUTCOMES:
systolic and diastolic blood pressure | Fifteen minutes after preparation for cesarean section
  mmHg
heart rate | Fifteen minutes after preparation for cesarean section
  beats per minute
body temperature | Fifteen minutes after preparation for cesarean section
  degrees Celsius
respiratory rate | Fifteen minutes after preparation for cesarean section
  beats per minute
fetal heart rate | Fifteen minutes after preparation for cesarean section
  beats per minute

CONTACTS AND LOCATIONS:
Locations (1):
- Neslihan Yılmaz Sezer, Ankara, Mamak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No